CLINICAL TRIAL: NCT06068166
Title: Thoracic Epidural Anesthesia Reduces Mortality and Rehospitalization for Patients With Heart Failure With Reduced Ejection Fraction：a Retrospective Matched Case-control Study
Brief Title: Thoracic Epidural Anesthesia Reduces Mortality and Rehospitalization for Patients With Heart Failure With Reduced Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEA
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Thoracic Epidural Anesthesia
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDMT plus TEA (Experimental): The patients received maximally tolerated guideline-directed medical therapy (GDMT) plus TEA.
  Thoracic epidural anesthesia (TEA), the infusion of anesthetic agents (eg, lidocaine or ropivacaine) into the epidural space, is used to achieve sympathetic block at the T1 to T4 levels in thoracic and abdominal surgical procedures.
  Interventions: Combination Product: TEA plus GDMT
- GDMT (Active Comparator): The patients received maximally tolerated GDMT.
  Interventions: Drug: GDMT

INTERVENTIONS:
Combination Product: TEA plus GDMT — Thoracic epidural anesthesia (TEA), the infusion of anesthetic agents (eg, lidocaine or ropivacaine) into the epidural space, is used to achieve sympathetic block at the T1 to T4 levels in thoracic and abdominal surgical procedures. Since 1995, Professor Liu Fengqi has pioneered the use of TEA to treat end-stage HFrEF and achieved surprising results. TEA could reduce the enlarged heart cavity, halt and reverse cardiac remodeling, and improve cardiac systolic and diastolic function. Currently, thousands of HFrEF patients have received TEA procedure. All the patients received maximally tolerated guideline-directed medical therapy (GDMT).
  Arms: GDMT plus TEA
Drug: GDMT — All the patients received maximally tolerated guideline-directed medical therapy (GDMT) alone.
  Arms: GDMT

SUMMARY:
Despite significant scientific breakthrough in management, patients with heart failure with reduced ejection fraction (HFrEF) remain high morbidity and mortality, with a 5-year survival rate of 25% after hospitalization for HFrEF. The autonomic nervous system (ANS), particularly the sympathetic nervous system (SNS), plays a critical compensatory role in maintaining cardiovascular homeostasis in the failing heart. This is critical given the huge unmet need for novel treatment strategies for HFrEF.

Thoracic epidural anesthesia (TEA), the infusion of anesthetic agents (eg, lidocaine or ropivacaine) into the epidural space, is used to achieve sympathetic block at the T1 to T4 levels in thoracic and abdominal surgical procedures. Since 1995, Professor Liu Fengqi has pioneered the use of TEA to treat end-stage HFrEF and achieved surprising results. TEA could reduce the enlarged heart cavity, halt and reverse cardiac remodeling, and improve cardiac systolic and diastolic function. Currently, thousands of HFrEF patients have received TEA procedure. However, it is unclear whether TEA could positively impact the clinical outcomes of patients with HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* The present study was a retrospective, observational, matched case-control study of 1,840 consecutive inpatients, in New York Heart Association functional class II-IV with a left ventricular ejection fraction (LVEF) ≤40%, who were hospitalized from July 2013 to August 2019.

Exclusion Criteria:

* Patients were excluded because of insufficient patient information, refusal to participate, or loss to follow-up by telephone. In patients with multiple hospitalizations during the time period, the first hospitalization was utilized in the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1840 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of heart failure mortality in the patients with HFrEF | 8.5 years
  Rate of heart failure mortality in the patients with HFrEF

SECONDARY OUTCOMES:
Rate of heart failure rehospitalization in the patients with HFrEF | 8.5 years
  Rate of heart failure rehospitalization in the patients with HFrEF